CLINICAL TRIAL: NCT01634048
Title: The Effect of Protein-enriched Diet on Body Composition and Appetite
Acronym: ProteinRich
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/LO/0592
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Overweight; Obese; Metabolic Syndrome; Non Alcoholic Fatty Liver Disease
Keywords: high protein diet; meal replacements; low calorie diet; intra hepatocellular lipid
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein low calorie meal replacements (Experimental): Meal replacements with added protein powder(1.34g pro/kg).
  Interventions: Dietary Supplement: High Protein, low calorie meal replacement
- Normal protein, low calorie meal replacement group (Sham Comparator): The control group will have standard meal replacements (0.8g protein/kg body weight).
  Interventions: Dietary Supplement: High Protein, low calorie meal replacement

INTERVENTIONS:
Dietary Supplement: High Protein, low calorie meal replacement — The high protein group will have meal replacements with added protein powder (to achieve 1.34g protein/kg body weight) and the control group will have standard meal replacements (0.8g protein/kg body weight). Meal replacements have been used in hundreds of previous human studies and are generally not found to be linked to any serious adverse effects.

SUMMARY:
Obesity is a major problem worldwide and current dietary interventions are not proving to be enough to cease the increase in levels of obesity and its detrimental side effects, such as nonalcoholic fatty liver disease (NAFLD).

Existing data suggests that adjustments in the macronutrient composition of the diet, more specifically the protein content, may have beneficial effects on body composition and an antiobesegenic effect on appetite. This may be important in terms of controlling body weight and reducing the amount of fatty tissue within our bodies and organs, and therefore preventing obesity and its health related side effects.

The investigators will perform a study to investigate whether a high protein low energy diet compared to a normal protein low energy diet, in overweight adults can modify appetite and aid loss of weight and fat mass. Subjects will receive either a high protein low energy diet (1.34g protein/kg body weight) or a normal protein low energy diet (0.8g protein/kg body weight) in the form of 2 meal replacements and one conventional meal per day with 2 snacks for 12 weeks.

HYPOTHESIS In overweight subjects with the metabolic syndrome, a 12 week dietary intervention with a high protein low energy diet will lead to a reduced appetite, body weight and fat mass, more specifically to a greater fall in levels of fat in the liver and pancreas than a low energy normal protein diet.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese people as classified by BMI 27-35kg/ m2 (inclusive)
* A Finnish Diabetes Risk Score (FINDRISC) >8 [22]
* Waist circumference measurement of ≥102cm in males or ≥88cm in females
* Assessed as appropriate for inclusion, based on a prestudy screening (see section 3.4)
* Willingness and ability to give written informed consent and willingness and ability to understand, to participate and to comply with the study requirements

Exclusion Criteria:

* Claustrophobia
* Pacemaker, metal implant, clips, implanted device, shrapnel or bullets, metal in eyes that precludes magnetic resonance imaging
* Treatment with any medication that might affect the study outcome (e.g., medication that is affecting appetite regulation and/or blood flow)
* Current pregnancy or breast feeding
* Delivery within the last year
* Bariatric surgery
* History of any disease with unknown outcome
* Significant intercurrent disease or history of clinically significant disease of any type, in particular liver, kidney, or heart disease, any form of diabetes mellitus or psychiatric illness (including Depression as defined by BDIII score above 28)
* History of cancer, excluding skin cancer
* History of severe or multiple allergies, severe adverse drug reaction or leucopenia
* Smokers
* Regular drinkers of more than three units of alcohol daily (1 unit = 300 ml beer, 1 glass wine, 1 measure spirit)
* Subjects who have had a fluctuation of body weight >5% in the 3 months prior to entering into the study
* History of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit
* Regular intake of overthecounter (OTC) medication (other than the occasional paracetamol/aspirin)
* Poor compliers or subjects unlikely to attend
* Blood donation within the 12 week period before the initial study dose

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Protein Low Calorie Meal Replacements | Normal Protein, Low Calorie Meal Replacement Group
Started | 21 | 18
Completed | 15 | 15
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Protein Low Calorie Meal Replacements | Normal Protein, Low Calorie Meal Replacement Group | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9) | 44 (14) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 12 | 23
  Asian | 3 | 3 | 6
  Mixed | 4 | 1 | 5
  Black | 1 | 2 | 3
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 21 | 18 | 39
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.6 (3.0) | 30.8 (2.4) | 30.7 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lipid Content of the Liver (Intrahepatocellular Lipid)
Description: Changes in body weight and body composition, more specifically visceral, muscle, liver and pancreas fat content will be measured using magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS). Individual's data will be compared at baseline and at 12 weeks of following the diet and also to that of the participants given normal protein low energy diets. This data may therefore support our hypothesis that high protein intakes may help to aid weight loss and reduce fat mass and would therefore be a viable option in the treatment of obesity.
Time Frame: Change from Baseline at 12 weeks
Measure: Mean (Standard Error); unit: % IHCL
Arm/Group | High Protein Low Calorie Meal Replacements | Normal Protein, Low Calorie Meal Replacement Group
Number analyzed (Participants) | 13 | 11
% IHCL
  IHCL Baseline | 27.9 (26.8) | 9.3 (5.6)
  IHCL 12 weeks | 21.4 (23.2) | 5.9 (5.0)
Statistical Analysis 1: Comparison: High Protein Low Calorie Meal Replacements vs Normal Protein, Low Calorie Meal Replacement Group; Test type: Superiority; p < 0.05, ANOVA

2. Secondary Outcome: Change in Appetite Regulation, Measured by VAS and Food Intake.
Description: It has also been suggested that highprotein diets are more beneficial in the regulation of appetite. We therefore aim to measure any changes in appetite whilst on a highprotein lowenergy diet compared to a normalprotein lowenergy diet. Changes in appetite will be measured using validated questionnaires assessing subjects feeling of hunger, pleasantness and volume able to eat as well as fullness. This data may support our hypothesis that highprotein intakes may alter appetite regulation and therefore be a useful in the treatment of obesity.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: kcal Energy
Arm/Group | High Protein Low Calorie Meal Replacements | Normal Protein, Low Calorie Meal Replacement Group
Number analyzed (Participants) | 10 | 12
kcal Energy
  Energy Intake Baseline | 1769 (205) | 1864 (156)
  Energy Intake 12 weeks | 1369 (125) | 1528 (114)

3. Other Pre Specified Outcome: Composite Appetite Score AUC (Area Under Curve)
Description: A composite appetite score was calculated combing all four appetite measures to give a summary measure of appetite. Each appetite measure was assessed using validated 100 mm visual analogue scales (VAS) for hunger, fullness, desire to eat, and prospective food consumption (PFC) with the most positive and most negative sensations anchoring opposite ends of the line, from 'Not at all' or 'Nothing' to 'Extremely' or 'A large amount'. Participants were asked to mark the line at the point corresponding to their perceived appetite at that time. There is no score which is better or worse.
  Composite Appetite score (mm min) = [desire to eat + hunger + (100 - fullness) + prospective consumption]/4, as described by (Anderson et al, 2002). This reflects the four appetite related VAS (visual analogue scale) questions and was used as a summary measure of appetite. Area Under the Curve (AUC) was calculated for composite appetites score using the trapezoidal rule. AUC scores range from 0-9000mm*min
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mm*min
Arm/Group | High Protein Low Calorie Meal Replacements | Normal Protein, Low Calorie Meal Replacement Group
Number analyzed (Participants) | 15 | 15
mm*min
  Composite Appetite Score (VAS) Baseline | 4063 (372) | 3376 (372)
  Composite Appetite Score (VAS) 12 weeks | 3728 (428) | 3370 (428)

ADVERSE EVENTS:
Arm/Group | High Protein Low Calorie Meal Replacements | Normal Protein, Low Calorie Meal Replacement Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes